CLINICAL TRIAL: NCT04294654
Title: Interventional, Open-label Study of Flexible Doses of Vortioxetine on Depressive Symptoms in Patients With Major Depressive Disorder and Early Dementia
Brief Title: Vortioxetine in Patients With Depression and Early Dementia
Acronym: MEMORY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18315A
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder; Dementia
MeSH Terms: conditions — Depressive Disorder, Major; Dementia | interventions — Vortioxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortioxetine (Experimental): 5 - 20 mg/day tablets
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine 5, 10 and 20 mg/day, tablets, orally Patients will receive 5 mg vortioxetine once daily for one week. At visit 3, the dose will be increased to 10 mg/day for all patients. Thereafter the dose may be adjusted to 5, 10 or 20 mg/day.

SUMMARY:
This study evaluates the effectiveness of vortioxetine on depressive symptoms in patients with depression and early dementia

ELIGIBILITY:
Inclusion Criteria:

* The patient has a primary diagnosis of recurrent Major Depressive Disorder (MDD) with onset before age of 55, diagnosed according to DSM-5®
* The current major depressive episode (MDE) must be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has had the current MDE for <6 months.
* The patient has a Montgomery and Åsberg Depression Rating Scale (MADRS) total score ≥26 at the Baseline Visit.
* The diagnosis of onset of dementia has occurred at least 6 months prior to screening and after already being diagnosed with MDD. The diagnosis of dementia must be documented in patient's medical records. When deemed necessary per investigator judgement of patient clinical status and early dementia, the patient must be accompanied by a caregiver to study visits.
* Patients with dementia associated with vitamin B12 or folate deficiency should not be enrolled.
* Patients with or without treatment for dementia can be enrolled. For patients on treatment for dementia, there must be no change in treatment during the study and patients must be on stable dose for at least 3 months prior to the Screening Visit.
* The patient has Mini Mental State Examination (MMSE) total score 20-24, inclusive.

Exclusion Criteria:

-The patient has any current psychiatric disorder or Axis I disorder (DSM-5® criteria), established as the primary diagnosis, other than MDD, as assessed using the Mini International Neuropsychiatric Interview (MINI) or another diagnostic interview.

Other in- and exclusion criteria may apply

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery and Åsberg Depression Rating Scale (MADRS) total score | from baseline to Week 12
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome.

SECONDARY OUTCOMES:
Change in Digit-Symbol Substitution Test (DSST) Substitution Test (DSST) score | from baseline to Week 12
  Digit Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning)."
Change in Rey Auditory Verbal Learning Test (RAVLT) score | from baseline to Week 12
  Rey Auditory Verbal Learning Task (RAVLT) is a cognitive test designed to assess verbal learning and memory, including immediate memory, efficiency of learning, retroactive and proactive interference effects, and encoding versus retrieval. It consists of a number of tasks, including immediate recall and delayed recall. The number of words correctly recalled on each task is recorded.
Change in Instrumental Activities of Daily Living (IADL) score | from baseline to Week 12
  The Instrumental Activities of Daily Living (IADL) measures an individual's ability to carry out tasks that are important for daily living and capture functional changes. Scores for each question range from 0 (no assistance needed) to 2 (full assistance needed), and are assessed by informant interview. The scores for IADL (0-14) is the outcome, with higher scores indicating lesser ability to carry out daily living tasks
Change in Clinical Global Impression - Severity (CGI-S) score | from baseline to Week 12
  The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Clinical Global Impression - Improvement (CGI-I) score | at Week 12
  The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Response defined by decrease in MADRS total score | At Week 12
  Response is defined as a 50% decrease from baseline in MADRS total score
Remission defined by MADRS score | at Week 12
  Remission is defined as MADRS ≤10
Change in Bath Assessment of Subjective Quality of Life in Dementia (BASQID) score | from baseline to Week 12
  The BASQID30 is a clinician rating scale designed to assess subjective quality of life (QoL) in patients with dementia. The BASQID contains 14 core questions, which are scored from 0 to 4, with 4 indicating a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (24):
- Marienthali Kliinik, Tallinn, Estonia
- France (2):
  - Cabinet du Docteur Karim Boutayeb, Viersat
  - Centre de Recherche-Hopital Geriatrique de Charpennes, Villeurbanne
- Italy (4):
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia, Province Of Brescia
  - Azienda Ospedaliera di Perugia - Policlinico Monteluce, Perugia, Umbria
  - Fondazione Universitaria G.D'Annunzio Ce.S.I. Centro Ricerca (Centro Scienze del l'Invecchiamento..., Chieti
  - Fondazione Santa Lucia IRCCS, Rome
- Poland (8):
  - Clinical Research Center Spolka z ograniczona odpowiedzialnoscia Medic-R Spolka Komandytowa, Poznan, Greater Poland Voivodeship
  - MlynowaMed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - NZOZ Dom Sue Ryder - Pallmed Sp. z o.o., Bydgoszcz
  - CareClinic, Katowice
  - Centrum Zdrowia Psychicznego Biomed - Jan Latala, Kielce
  - Niepubliczny Zaklad Opieki Psychiatrycznej Mentis, Leszno
  - Centrum Medyczne Luxmed Sp.Z O.O., Lublin
  - Nzoz Syntonia, Pruszcz Gdański
- South Korea (5):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - University Clinical Hospital of Valladolid, Valladolid
  - Hospital Río Hortega, Valladolid
  - Centro de Saude de Lavadores, Vigo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christensen MC, Schmidt SN, Grande I. Effectiveness of vortioxetine in patients with major depressive disorder and early-stage dementia: The MEMORY study. J Affect Disord. 2023 Oct 1;338:423-431. doi: 10.1016/j.jad.2023.06.024. Epub 2023 Jun 12. PMID 37315590